CLINICAL TRIAL: NCT04623346
Title: Orthopaedic Conservative Treatment in the Time of Covid-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Bulent KARSLIOGLU, Orthopedics and Traumatology specialist, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: Treatment in the time of Covid
Record Dates: First submitted 2020-11-07; First posted 2020-11-10 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Ankle Fractures; Proximal Humeral Fracture; Wrist Fracture
MeSH Terms: conditions — Ankle Fractures; Shoulder Fractures; Wrist Fractures | interventions — Observation; Surgical Procedures, Operative; Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Weber B-type Ankle fractures in prepandemic period: Patients with AO Weber B-type ankle fracture in prepandemic period
- Weber B-type Ankle fractures in pandemic period: Patients with AO Weber B-type ankle fracture in pandemic period
  Interventions: Procedure: Observation for study group
- Wrist fractures in prepandemic period: Patients with extraarticular distal radius fracture in prepandemic period
- Wrist fractures in pandemic period: Patients with extraarticular distal radius fracture in pandemic period
  Interventions: Procedure: Observation for study group
- Proximal humerus fractures in prepandemic period: Patients with 2-part,3-part and 4-part fractures in prepandemic period
- Proximal humerus fractures in pandemic period: Patients with 2-part,3-part and 4-part fractures in pandemic period
  Interventions: Procedure: Observation for study group

INTERVENTIONS:
Procedure: Observation for study group — Patients with Weber B-type Ankle fractures, extraarticular wrist fractures and proximal humerus fractures were followed with conservative manner( cast or sling)
  Other Names: Surgery for control group
  Groups: Proximal humerus fractures in pandemic period; Weber B-type Ankle fractures in pandemic period; Wrist fractures in pandemic period

SUMMARY:
This is a one centered retrospective study. Tendency for surgical interventions in the pre-pandemic period was reduced to protect surgical team and patients. The investigators aimed to find out the answer to the following question: will conservative treatment be the shining star in the post pandemic period?

DETAILED DESCRIPTION:
The researchers compared the treatments performed for fractures during the Covid 19 pandemic period with the treatments performed in the prepandemic period. For this purpose, they tried to measure the effectiveness of the treatments according to clinical scoring by forming 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with extraarticular distal radius fracture, proximal humerus fracture and Weber type B ankle fracture were treated conservatively during March 11, 2020 and 11 August, 2020

Exclusion Criteria:

* Surgically treated patients during March 11, 2020 and 11 August, 2020

Min Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who admitted to emergency orthopedics department between March 11, 2020 and August 11, 2020
Sampling Method: Probability Sample
Enrollment: 262 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the two groups in terms of bony union | 12 week
  The investigators aimed to investigate the duration of bone union time between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- SBU Prof. Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Holshue ML, DeBolt C, Lindquist S, Lofy KH, Wiesman J, Bruce H, Spitters C, Ericson K, Wilkerson S, Tural A, Diaz G, Cohn A, Fox L, Patel A, Gerber SI, Kim L, Tong S, Lu X, Lindstrom S, Pallansch MA, Weldon WC, Biggs HM, Uyeki TM, Pillai SK; Washington State 2019-nCoV Case Investigation Team. First Case of 2019 Novel Coronavirus in the United States. N Engl J Med. 2020 Mar 5;382(10):929-936. doi: 10.1056/NEJMoa2001191. Epub 2020 Jan 31. PMID 32004427
- [Background] Chen YC, Lin WC. Risk of long-term infection-related death in clinical osteoporotic vertebral fractures: A hospital-based analysis. PLoS One. 2017 Aug 9;12(8):e0182614. doi: 10.1371/journal.pone.0182614. eCollection 2017. PMID 28793342
- [Background] Mi B, Xiong Y, Lin Z, Panayi AC, Chen L, Liu G. COVID-19 Orthopaedic Safe Care Toolset: Guidelines for the Diagnosis and Management of Patients with Fracture and COVID-19. J Bone Joint Surg Am. 2020 Jul 1;102(13):1116-1122. doi: 10.2106/JBJS.20.00532. PMID 32618909
- [Background] Guo X, Wang J, Hu D, Wu L, Gu L, Wang Y, Zhao J, Zeng L, Zhang J, Wu Y. Survey of COVID-19 Disease Among Orthopaedic Surgeons in Wuhan, People's Republic of China. J Bone Joint Surg Am. 2020 May 20;102(10):847-854. doi: 10.2106/JBJS.20.00417. PMID 32271208
- [Background] Saxena A, Bullock M, Danoff JR, Rodd DS, Fischer SJ, Stronach BM, Levine BR. Educating Surgeons to Educate Patients About the COVID-19 Pandemic. J Arthroplasty. 2020 Jul;35(7S):S65-S67. doi: 10.1016/j.arth.2020.04.037. Epub 2020 Apr 18. PMID 32340829
- [Background] Lei S, Jiang F, Su W, Chen C, Chen J, Mei W, Zhan LY, Jia Y, Zhang L, Liu D, Xia ZY, Xia Z. Clinical characteristics and outcomes of patients undergoing surgeries during the incubation period of COVID-19 infection. EClinicalMedicine. 2020 Apr 5;21:100331. doi: 10.1016/j.eclinm.2020.100331. eCollection 2020 Apr. PMID 32292899
- [Background] Handoll HH, Keding A, Corbacho B, Brealey SD, Hewitt C, Rangan A. Five-year follow-up results of the PROFHER trial comparing operative and non-operative treatment of adults with a displaced fracture of the proximal humerus. Bone Joint J. 2017 Mar;99-B(3):383-392. doi: 10.1302/0301-620X.99B3.BJJ-2016-1028. PMID 28249980
- [Background] Orman S, Mohamadi A, Serino J, Murphy J, Hanna P, Weaver MJ, Dyer G, Nazarian A, von Keudell A. Comparison of surgical and non-surgical treatments for 3- and 4-part proximal humerus fractures: A network meta-analysis. Shoulder Elbow. 2020 Apr;12(2):99-108. doi: 10.1177/1758573219831506. Epub 2019 Feb 28. PMID 32313559
- [Background] Maier D, Jaeger M, Izadpanah K, Strohm PC, Suedkamp NP. Proximal humeral fracture treatment in adults. J Bone Joint Surg Am. 2014 Feb 5;96(3):251-61. doi: 10.2106/JBJS.L.01293. PMID 24500588
- [Background] Hertel R, Hempfing A, Stiehler M, Leunig M. Predictors of humeral head ischemia after intracapsular fracture of the proximal humerus. J Shoulder Elbow Surg. 2004 Jul-Aug;13(4):427-33. doi: 10.1016/j.jse.2004.01.034. PMID 15220884
- [Background] Murray IR, Amin AK, White TO, Robinson CM. Proximal humeral fractures: current concepts in classification, treatment and outcomes. J Bone Joint Surg Br. 2011 Jan;93(1):1-11. doi: 10.1302/0301-620X.93B1.25702. PMID 21196536
- [Background] Martin AG. Weber B ankle fracture: an unnecessary fracture clinic burden. Injury. 2004 Aug;35(8):805-8. doi: 10.1016/j.injury.2003.12.013. PMID 15246805
- [Background] Mittal R, Harris IA, Adie S, Naylor JM; CROSSBAT Study Group. Surgery for Type B Ankle Fracture Treatment: a Combined Randomised and Observational Study (CROSSBAT). BMJ Open. 2017 Mar 27;7(3):e013298. doi: 10.1136/bmjopen-2016-013298. PMID 28348185
- [Background] Van Schie-Van der Weert EM, Van Lieshout EM, De Vries MR, Van der Elst M, Schepers T. Determinants of outcome in operatively and non-operatively treated Weber-B ankle fractures. Arch Orthop Trauma Surg. 2012 Feb;132(2):257-63. doi: 10.1007/s00402-011-1397-z. Epub 2011 Sep 30. PMID 21959696
- [Background] Young BT, Rayan GM. Outcome following nonoperative treatment of displaced distal radius fractures in low-demand patients older than 60 years. J Hand Surg Am. 2000 Jan;25(1):19-28. doi: 10.1053/jhsu.2000.jhsu025a0019. PMID 10642469
- [Background] Chang HC, Tay SC, Chan BK, Low CO. Conservative treatment of redisplaced Colles' fractures in elderly patients older than 60 years old - anatomical and functional outcome. Hand Surg. 2001 Dec;6(2):137-44. doi: 10.1142/s0218810401000606. PMID 11901459
- [Background] Fujii K, Henmi T, Kanematsu Y, Mishiro T, Sakai T, Terai T. Fractures of the distal end of radius in elderly patients: a comparative study of anatomical and functional results. J Orthop Surg (Hong Kong). 2002 Jun;10(1):9-15. doi: 10.1177/230949900201000103. PMID 12401915
- [Background] Anzarut A, Johnson JA, Rowe BH, Lambert RG, Blitz S, Majumdar SR. Radiologic and patient-reported functional outcomes in an elderly cohort with conservatively treated distal radius fractures. J Hand Surg Am. 2004 Nov;29(6):1121-7. doi: 10.1016/j.jhsa.2004.07.002. PMID 15576226